CLINICAL TRIAL: NCT02689986
Title: The CAD5 Study::Therapy for Chronic Cold Agglutinin Disease: A Prospective, Non-randomized International Multicenter Trial on the Safety and Efficacy of Bendamustine and Rituximab Combination Therapy
Brief Title: Bendamustine and Rituximab Combination Therapy for Cold Agglutinin Disease
Acronym: CAD5
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helse Fonna (Other)
Responsible Party: Principal Investigator, Sigbjorn Berentsen, MD, PhD, Helse Fonna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAD5
Record Dates: First submitted 2016-02-16; First posted 2016-02-24 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Cold Agglutinin Disease; Autoimmune Hemolytic Anemia
Keywords: Cold agglutinin; Cold agglutinin disease; Anemia; Hemolytic; Autoimmune; Bendamustine; Rituximab
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune; Anemia; Hemolysis | interventions — Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment arm (Experimental): Bendamustine, Rituximab
  Interventions: Drug: Bendamustine, Rituximab

INTERVENTIONS:
Drug: Bendamustine, Rituximab — Bendamustine, Rituximab
  Other Names: Levact, MabThera

SUMMARY:
Prospective, non-randomized multicenter study on the safety and efficacy of combination therapy with bendamustine and rituximab for chronic cold agglutinin disease.

DETAILED DESCRIPTION:
Background

Chronic cold agglutinin disease (CAD) is mediated by monoclonal cold-reactive autoantibodies that bind to erythrocyte surface antigens, causing hemagglutination and complement-mediated hemolysis. Anemia is severe in one-third of patients (hemoglobin level 8.0 g/dL or lower). Cold-induced circulatory symptoms are present in more than 90% of patients and may be disabling. CAD not associated with overt lymphoma or other disease has traditionally been classified as primary or idiopathic. A monoclonal lymphoproliferative bone marrow disorder can, however, be demonstrated by flow cytometry in 90% and by histology in approximately 75% of these patients, characterized by clonal proliferation of CD20+, kappa+ B-cells.

Approximately two-thirds of the patients experience exacerbation during febrile illnesses. During steady-state CAD, a majority of patients have low levels of complement proteins C3 and C4 because of a continuous consumption. These low levels, in particular low C4 availability, seem to be rate-limiting for hemolysis and prevent full-blown activation of the complement cascade with C5 cleavage and intravascular hemolysis. During acute phase reaction, C3 and C4 levels increase due to an enhanced production, resulting in exacerbation of hemolysis.

Counseling on cold avoidance has been recommended as the treatment of choice for most patients with primary CAD. A systematic review showed, however, that in more than 70% of cases, the physician and/or the patient did not perceive such measures as sufficient). Many standard therapies used in other autoimmune diseases or indolent lymphomas are inefficient, e.g. corticosteroids, alkylating agents, interferon-α and, probably, purine analogue single agent therapy. Treatment with the chimeric monoclonal anti-CD20 antibody rituximab has been shown in prospective studies to induce remission in more than half of patients. Almost all responses were partial, and the median response duration was less than one year. In a subsequent, prospective non-randomized trial of fludarabine and rituximab combination therapy in 29 patients, 22 patients (76%) responded, 6 (21%) achieving CR and 16 (55%) achieving PR. Among 10 patients non-responsive to rituximab monotherapy, CR was observed after the combination therapy in one patient and PR in six. Median increase in Hb level was 3.1 g/dL in the responders and 4.0 g/dL among those who achieved CR. Median time to response was 4.0 months. Lower quartile of response duration was not reached after 33 months, and estimated median response duration was more than 66 months. Targeting the pathogenic B-cell clone efficiently seems important for the achievement of remission.

Though the rituximab-based therapies have been a first major achievement in therapy for CAD, some problems remain to be solved. First, a considerable number of patients do not respond to rituximab monotherapy. Second, although the use of fludarabine and rituximab in combination has resulted in high response rates and prolonged response duration, toxicity is significant and there are still some non-responders. Third, the therapeutic approaches should probably be individualized; e.g., fludarabine therapy may bring about problems in the younger patients because of late-occurring adverse events and in the older ones because of short-term hematologic toxicity.

The antineoplastic drug, bendamustine hydrochloride, combines the 2-chlorethylamine group of the nitrogen mustard derived alkylating agents with the benzimidazole ring structures of the purine analogue. Bendamustine has been shown to be highly active in a variety of lymphoproliferative disorders. The combination of bendamustine and rituximab has produced high overall and complete response rates and prolonged remissions with only moderate and manageable toxicity in Waldenström's macroglobulinemia, which is closely related to primary CAD. In an attempt to improve on the therapeutic efficacy achieved with the rituximab-based regimens and the toxicity profile of the fludarabine-rituximab combination, the investigators want to study the safety and efficacy of bendamustine and rituximab combination therapy in patients with primary CAD.

Clinical study

The study is a prospective, non-randomized multicenter trial designed to investigate the efficacy and safety of bendamustine and rituximab combination therapy in patients with CAD requiring treatment.

Because of the low prevalence of CAD, it will be unrealistic to undertake a statistically robust randomized study. The investigators aim to include 50 patients during a study period of three years.

2.1 Study objective

The objective is to assess safety and efficacy of combination therapy with bendamustine and rituximab in patients with CAD.

Primary endpoints: Rate of complete and partial responses, respectively. Secondary endpoints: Time to response; time to best response; hematological toxicity grade 4; frequency of dose reduction; response duration.

2.2. Ethics

The trial will be carried out in accordance with the Helsinki Declaration and the current statutory requirements and legislation in the participating countries. The study has been approved by the relevant Medical Research Ethics Committees, the Norwegian Medicines Agency and the relevant regulatory authorities of each participating country. Data will be recorded anonymously, but a numeric code will be assigned in order to be able to track the data. All investigators as well as the ethics committees and relevant health authorities, however, will have access to the source data. The principal investigator in each country will establish monitoring of the study by an independent monitor as required.

2.3 Study design

Prospective, non-randomized international multicenter study.

2.4 Study population

In principle, individuals aged at least 18 years can be included, although enrollment of patients younger than 40 years is unlikely due to the age-specific prevalence of the disease.

3 The drugs

3.1 Rituximab

Rituximab is a humanized, chimeric monoclonal anti-CD20 antibody. Treatment with rituximab is considered an established, not experimental therapy for CAD, and involved physicians and nurses should be familiar with its administration, therapeutic and adverse effects and safety issues. In particular, they should be able to identify and manage any infusion-related side effects.

3.2 Bendamustine

Bendamustine is the experimental drug of this trial, marketed by Mundipharma/Norpharma. The drug is approved in the participating countries for the treatment of non-Hodgkin's lymphoma, chronic lymphocytic leukemia and multiple myeloma. It is a cytotoxic agent combining the 2-chlorethylamine group of the nitrogen mustard derived alkylating agents with the benzimidazole ring structures of the purine nucleoside analogues. Precautions and warnings include the possibility of myelosuppression, infections, skin reactions, caution in patients with cardiac disorders, nausea, vomiting, tumor lysis syndrome (very unlikely in primary CAD), anaphylaxis and extravasation.

4 Inclusion of patients.

Examination at inclusion

4.1 History.

Clinical and radiological examination Year of first occurrence of clinical symptoms is registered along with data on hemolytic anemia, circulatory symptoms, cold- or fever-induced exacerbation, previous therapies, lymph node enlargement and spleen enlargement (clinical assessment). Chest radiograph and abdominal ultrasonography should be done if not already performed during the last four months.

4.2 Blood tests

Hemolysis is detected and quantified based on Hb, MCV, reticulocyte count (x 109/L), LDH, bilirubin and haptoglobin. These measurements should be done twice during the last two months before treatment.

Hematological, biochemical and immunological assessments should be done once at inclusion + 2 weeks:

* WBC, leukocyte differential count, platelet count
* Iron, transferrin (or TIBC), ferritin, cobalamine and folate
* CRP
* Quantification of IgM, IgG and IgA Serum electrophoresis for detection and identification of monoclonal immunoglobulins (including immunofixation when appropriate)
* Cold agglutinin titer
* Specific direct antiglobulin test (DAT, direct Coombs' test), i.e. using polyspecific antiserum, anti-C3d and anti-IgG)
* Complement assessments (C3 and C4)
* CMV and VZV antibodies
* Serological tests for hepatitis B and C
* Freezing of 5 ml EDTA-blood for possible later DNA-based studies

  5 Therapy

Treatment schedule Day 1: Rituximab; 375 mg/m2 Day 1-2: Bendamustine; dosage: see Section 5.2 Day 29: Rituximab; 375 mg/m2 Day 29-30: Bendamustine; dosage: see Section 5.2 and 5.4 Day 57: Rituximab; 375 mg/m2 Day 57-58: Bendamustine; dosage: see Section 5.2 and 5.4 Day 85: Rituximab; 375 mg/m2 Day 85-86: Bendamustine; dosage: see Section 5.2 and 5.4 5.2 Initial bendamustine dose Patients with no previous cytotoxic therapy and no history of myelosuppression receive bendamustin at an initial dose of 90 mg/m2 day 1 and 2 (dose level A).

In patients who have been previously treated with a fludarabine-containing regimen, the initial bendamustine dose is 70 mg/m2 day 1 and 2 (dose level B).

In patients who have previously received myelosuppressive agents other than purine analogues, the choice of initial dose level A or B is based on an individualized assessment.

Bendamustine solution for infusion should be prepared according to the manufacturer's recommendations. The solution should be administered by intravenous infusion over 60 minutes. Antiemetic prophylaxis is given according to local routines or based on an individualized assessment.

Rituximab should be administered according to the manufacturer's recommendations and the routines of the participating hospital. Rapid (90 minutes) infusion is allowed during cycle 2-4 provided there has been no infusion-related adverse event during the preceding rituximab infusion.

For drug stability reasons, an in-line blood warmer should not be used for the infusion of bendamustine or rituximab. The infusion solution should have room temperature; and the patient, in particular the extremity chosen for infusion, should be kept warm during the procedure.

Dose adjustments

In case of significant toxicity, the dose of bendamustine should be reduced as specified by protocol. Any adverse event should be recorded in the appropriate CRF. For reporting of SAEs and SUSARs, see Protocol

6 Follow-up

6.1 Follow-up first 6 months after therapy

A) The following measurements must be done monthly during the first six months after the last cycle of any combination therapy:

I) All measurements listed in Paragraph 6.1.B.

II) In case of reduction of a previously elevated IgM level to the normal range, serum electrophoresis and immunofixation should be performed at the next visit.

III) Number of blood transfusions after the previous monthly visit. B.) At the fourth monthly visit after completion of the last combination therapy cycle, bone marrow biopsy and flow cytometric immunophenotyping of bone marrow aspirate are performed.

ELIGIBILITY:
Inclusion Criteria:

1. CAD diagnosis defined by the combination of -

   1. Chronic hemolysis
   2. Cold agglutinin titer 64 or higher
   3. Positive direct antiglobulin test when performed with polyspecific antiserum, negative (or only weakly positive) with anti-IgG, and strongly positive with anti-C3d
2. The presence of a clonal B-cell lymphoproliferative disorder defined by -

   1. Monoclonal band by serum electrophoresis with immunofixation, and/or
   2. CD20 positive lymphocyte population with cellular kappa/lamda-ratio higher than 3.5 or less than 0.9, using flowcytometric immunophenotyping of bone marrow aspirates
3. Indication for therapy, i.e. significant anemia and/or considerable cold-induced circulatory symptoms
4. Written informed consent

Exclusion Criteria:

1. An aggressive lymphoma
2. Non-lymphatic malignant disease other than basal cell carcinoma of the skin. A history of probably cured cancer is not an exclusion criterion.
3. Known HIV infection
4. Acute or chronic hepatitis B or C
5. Liver failure or active parenchymal liver disease. Bilirubin levels higher than 51 mol/L (3.0 mg/dL) when due to hepatic impairment. Elevated serum bilirubin level due to hemolysis is not an exclusion criterion.
6. Pregnancy or breast-feeding
7. Patients of childbearing age who are not willing to use safe contraception during the entire study period and 6 months following its cessation
8. All contraindications to the study drugs will be regarded as exclusion criteria.
9. Age below 18 years
10. Inability to cooperate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Frequency of complete and partial responses (CR/PR) | 6 months
  Responses will be assessed using the following, previously published definitions:
  Complete response (CR), Absence of anemia, no signs of hemolysis, no clinical symptoms of CAD, undetectable serum monoclonal protein, and no signs of clonal lymphoproliferation by bone marrow histology, immunohistochemistry and flow cytometry.
  Partial response (PR), Stable increase in hemoglobin levels by at least 2.0 g/dL or to the normal range, combined with a reduction of serum IgM concentrations by at least 50% or to the normal range, improvement of clinical symptoms, and transfusion independency.
  Non-response (NR), Patients not meeting the criteria for CR or PR.

SECONDARY OUTCOMES:
Time to response (TTR) | 6 months
  Time to response (TTR) is the time from start of therapy to the achievement of any degree of response.
Time to best response (TTBR) | 1 year
  Time to best response (TTBR) is the time from start of therapy to the observation of the highest hemoglobin level achieved + 0.5 g/dL.
Response duration | Through study completion; an average of 2 years
  Response duration is the time from achievement of any degree of response to relapse. Relapse is defined by one or more of the following events: A decline in hemoglobin level by at least 2.0 g/dL from the highest level achieved or to below 10.0 g/dL; transfusion requirement; or recurrence of significant cold-induced circulatory symptoms.
Number of participants with treatment-related adverse events as assessed by current CTCAE criteria | Through study completion; an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sigbjorn Berentsen, MD, PhD, Study Chair — Department of Research and Innovation, Haugesund Hospital; Markku Oksman, MD, Principal Investigator — Turku University Hospital, Turku, Finland; Henrik Birgens, MD, PhD, Principal Investigator — Herlev University Hospital, Copenhagen, Denmark; Geir E Tjonnfjord, MD, PhD, Principal Investigator — Oslo University Hospital, Oslo, Norway
Locations (8):
- Herlev University Hospital, Copenhagen, Denmark
- Turku University Hospital, Turku, Finland
- Norway (6):
  - Haukeland University Hospital, Bergen
  - Vestre Viken Hospital, Drammen
  - Haugesund Hospital, Haugesund
  - Akershus University Hospital, Nordbyhagen
  - Oslo University Hospital, Oslo
  - St Olav University Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: Yes
Data are to be shared between authors before final analysis and publication.

REFERENCES:
- [Background] Michel M. Classification and therapeutic approaches in autoimmune hemolytic anemia: an update. Expert Rev Hematol. 2011 Dec;4(6):607-18. doi: 10.1586/ehm.11.60. PMID 22077525
- [Background] Randen U, Troen G, Tierens A, Steen C, Warsame A, Beiske K, Tjonnfjord GE, Berentsen S, Delabie J. Primary cold agglutinin-associated lymphoproliferative disease: a B-cell lymphoma of the bone marrow distinct from lymphoplasmacytic lymphoma. Haematologica. 2014 Mar;99(3):497-504. doi: 10.3324/haematol.2013.091702. Epub 2013 Oct 18. PMID 24143001
- [Background] Berentsen S, Tjonnfjord GE. Diagnosis and treatment of cold agglutinin mediated autoimmune hemolytic anemia. Blood Rev. 2012 May;26(3):107-15. doi: 10.1016/j.blre.2012.01.002. Epub 2012 Feb 12. PMID 22330255
- [Background] Berentsen S, Randen U, Vagan AM, Hjorth-Hansen H, Vik A, Dalgaard J, Jacobsen EM, Thoresen AS, Beiske K, Tjonnfjord GE. High response rate and durable remissions following fludarabine and rituximab combination therapy for chronic cold agglutinin disease. Blood. 2010 Oct 28;116(17):3180-4. doi: 10.1182/blood-2010-06-288647. Epub 2010 Jul 15. PMID 20634373
- [Background] Berentsen S, Beiske K, Tjonnfjord GE. Primary chronic cold agglutinin disease: an update on pathogenesis, clinical features and therapy. Hematology. 2007 Oct;12(5):361-70. doi: 10.1080/10245330701445392. PMID 17891600
- [Background] Berentsen S, Ulvestad E, Langholm R, Beiske K, Hjorth-Hansen H, Ghanima W, Sorbo JH, Tjonnfjord GE. Primary chronic cold agglutinin disease: a population based clinical study of 86 patients. Haematologica. 2006 Apr;91(4):460-6. PMID 16585012
- [Background] Berentsen S, Ulvestad E, Gjertsen BT, Hjorth-Hansen H, Langholm R, Knutsen H, Ghanima W, Shammas FV, Tjonnfjord GE. Rituximab for primary chronic cold agglutinin disease: a prospective study of 37 courses of therapy in 27 patients. Blood. 2004 Apr 15;103(8):2925-8. doi: 10.1182/blood-2003-10-3597. Epub 2003 Dec 30. PMID 15070665
- [Background] Schollkopf C, Kjeldsen L, Bjerrum OW, Mourits-Andersen HT, Nielsen JL, Christensen BE, Jensen BA, Pedersen BB, Taaning EB, Klausen TW, Birgens H. Rituximab in chronic cold agglutinin disease: a prospective study of 20 patients. Leuk Lymphoma. 2006 Feb;47(2):253-60. doi: 10.1080/10428190500286481. PMID 16321854
- [Background] Gueli A, Gottardi D, Hu H, Ricca I, De Crescenzo A, Tarella C. Efficacy of rituximab-bendamustine in cold agglutinin haemolytic anaemia refractory to previous chemo-immunotherapy: a case report. Blood Transfus. 2013 Apr;11(2):311-4. doi: 10.2450/2012.0166-12. Epub 2013 Jan 22. No abstract available. PMID 23399352
- [Background] Berentsen S, Ulvestad E, Tjonnfjord GE. B-lymphocytes as targets for therapy in chronic cold agglutinin disease. Cardiovasc Hematol Disord Drug Targets. 2007 Sep;7(3):219-27. doi: 10.2174/187152907781745279. PMID 17896962
- [Background] Ulvestad E, Berentsen S, Bo K, Shammas FV. Clinical immunology of chronic cold agglutinin disease. Eur J Haematol. 1999 Oct;63(4):259-66. doi: 10.1111/j.1600-0609.1999.tb01887.x. PMID 10530415
- [Background] Ulvestad E, Berentsen S, Mollnes TE. Acute phase haemolysis in chronic cold agglutinin disease. Scand J Immunol. 2001 Jul-Aug;54(1-2):239-42. doi: 10.1046/j.1365-3083.2001.00960.x. PMID 11439172
- [Background] Berentsen S. How I manage cold agglutinin disease. Br J Haematol. 2011 May;153(3):309-17. doi: 10.1111/j.1365-2141.2011.08643.x. Epub 2011 Mar 8. PMID 21385173
- [Background] Swiecicki PL, Hegerova LT, Gertz MA. Cold agglutinin disease. Blood. 2013 Aug 15;122(7):1114-21. doi: 10.1182/blood-2013-02-474437. Epub 2013 Jun 11. PMID 23757733
- [Background] Stone MJ. Heating up cold agglutinins. Blood. 2010 Oct 28;116(17):3119-20. doi: 10.1182/blood-2010-07-297523. PMID 21030565
- [Background] Berentsen S, Tjonnfjord GE, Shammas FV, Bergheim J, Hammerstrom J, Langholm R, Ulvestad E. No response to cladribine in five patients with chronic cold agglutinin disease. Eur J Haematol. 2000 Jul;65(1):88-90. doi: 10.1034/j.1600-0609.2000.9l201.x. No abstract available. PMID 10914950
- [Background] Rummel M, Kaiser U, Balser C, Stauch M, Brugger W, Welslau M, Niederle N, Losem C, Boeck HP, Weidmann E, von Gruenhagen U, Mueller L, Sandherr M, Hahn L, Vereshchagina J, Kauff F, Blau W, Hinke A, Barth J; Study Group Indolent Lymphomas. Bendamustine plus rituximab versus fludarabine plus rituximab for patients with relapsed indolent and mantle-cell lymphomas: a multicentre, randomised, open-label, non-inferiority phase 3 trial. Lancet Oncol. 2016 Jan;17(1):57-66. doi: 10.1016/S1470-2045(15)00447-7. Epub 2015 Dec 5. PMID 26655425
- [Derived] Berentsen S, Randen U, Oksman M, Birgens H, Tvedt THA, Dalgaard J, Galteland E, Haukas E, Brudevold R, Sorbo JH, Naess IA, Malecka A, Tjonnfjord GE. Bendamustine plus rituximab for chronic cold agglutinin disease: results of a Nordic prospective multicenter trial. Blood. 2017 Jul 27;130(4):537-541. doi: 10.1182/blood-2017-04-778175. Epub 2017 May 22. PMID 28533306